CLINICAL TRIAL: NCT05867784
Title: Effect of Vitamin D Supplementation on the Efficacy of Ustekinumab in the Treatment of Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2023-01-203
Record Dates: First submitted 2023-05-10; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Ustekinumab; Vitamin D Supplementation; Crohn's Disease; Clinical Efficacy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- supplementary group: take vitamin D supplementation (400 IU/day) during VDZ treatment
- non-supplementary group: not take vitamin D supplementation (400 IU/day) during VDZ treatment

SUMMARY:
It is uncertain whether vitD3 supplementation is beneficial for the remission of Crohn's disease (CD). The effects of vitD3 supplements on the efficacy of ustekinumab in Chinese CD patients were retrospectively analyzed. Methods: Patients with moderate to severe CD were recorded. These patients were initially treated with UST. VitD3 supplementation was defined as 400IU/d vitD3 supplementation during the first infusion of UST and continued throughout the follow-up period. Disease activity was assessed using Harvey Bradshaw Index.

ELIGIBILITY:
Inclusion Criteria:

* moderate-to-severe CD
* Treated with Ustekinumab

Exclusion Criteria:

* had recent supplementation of vitD3
* pregnant
* had cognitive/developmental disorders that affected their ability to complete the study procedures
* had medical illness or therapies potentially affecting bone, nutrition or growth status
* unknown or untested baseline serum 25(OH)D level

Ages: 15 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Chinese
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Serum 25 (OH) D level | 24 weeks
  Vitamin D deficiency is defined as serum 25 (OH) D level<20 μ g/L
disease activity | 24weeks
  Harvey Bradshaw Index，mild: 0 to 8, moderate: 9 to 16, severe: 17 to 25

SECONDARY OUTCOMES:
Serum 25 (OH) D level | 8 weeks
  Vitamin D deficiency is defined as serum 25 (OH) D level<20 μ g/L

CONTACTS AND LOCATIONS:
Overall Officials: Yi Jiang, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- SAHWenzhouMU, Wenzhou, Zhejiang, China